CLINICAL TRIAL: NCT01847846
Title: Analysis of a New CPAP Mask for Patients With Sleep-disordered Breathing and Treated With Positive Airway Pressure (PAP) Thearapy
Brief Title: Analysis of a New Mask for Positive Airway Pressure (PAP) Device Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MA07052013; MA07052013 (Other: Clinical Trial Notification (CTN) scheme, Therapeutic Goods Act (TGA), Australia)
Record Dates: First submitted 2013-04-30; First posted 2013-05-07 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: CPAP; mask; microorganisms
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prototype mask (Experimental): Participants will be randomised to trial the new prototype mask for 4 and 8 weeks. The prototype mask will be used in conjunction with the participant's home CPAP machine. The participant's will be instructed to use the prototype mask every night until the completion of the trial. No changes will be made to the participant's prescribed CPAP settings.
  Interventions: Device: CPAP mask - prototype

INTERVENTIONS:
Device: CPAP mask - prototype — prototype mask, wore for all sleeps for 4 and 8 weeks (as randomly selected). Mask to be used in conjunction with participant's usual prescribed CPAP settings.
  Other Names: PAP mask

SUMMARY:
BACKGROUND AND AIMS Continuous positive airway pressure (CPAP) is an effective therapy to treat sleep apnea. Sleep apnea is a condition where the airways collapse when the patient is asleep. CPAP treats sleep apnea by delivering an air pressure to the airways, splinting the airways open. CPAP is a device that sits besides the bed and is applied to the patient using a face mask.

The development of new CPAP masks is an on-going focus at ResMed Ltd in a bid to improve comfort and user compliance. ResMed are developing a new mask and investigations are required to evaluate mask performance over time.

ResMed Ltd design and manufacturer CPAP masks. The revision and development of masks is an on-going focus of the company in a bid to improve usability and patient compliance while maintaining optimum treatment. ResMed is developing a new mask. Investigations are therefore required to determine how much matter is built-up on the mask over time and to evaluate mask performance (including comfort and seal) and efficacy.

AIMS

The aims of the study are:

1. To measure and compare the change in the abundance of microbes on the new mask over a period of 8 weeks
2. To measure and compare the change in comfort, seal, stability, efficacy, leak and user compliance of this new mask over a period of 8 weeks
3. To measure and compare the change in comfort, seal, stability, efficacy, leak and user compliance of this new mask versus an available mask

It is hypothesised that:

1. The new mask acquires microbes from the user but there is no difference in the abundance of microorganisms between 2 and 8 weeks.
2. The new mask maintains the same degree of comfort, seal, stability, efficacy, leak and compliance between 2 and 8 weeks.
3. Compared to the existing mask, the new mask provides a higher degree of comfort, seal and stability and improves user compliance. The new mask also maintains efficacy, and maintains or reduces leak compared to the current masks.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 yrs old
* Diagnosed with obstructive sleep apnoea
* Been using CPAP therapy for at least 6 months

Exclusion Criteria:

* Has a lung disease/condition
* Using bilevel therapy
* Is unable to participate for the duration of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
To measure and compare the prevalence of microorganisms within the new mask over a period of 8 weeks | up to 8 weeks of use
  The mask is for single user use only. The participants will be instructed not to wash or clean the material for the duration of the study. The mask will be returned in a sealed bag and sent off for testing within 24 hrs after the trial.

SECONDARY OUTCOMES:
Measure and compare mask efficacy over a period of 8 weeks | After 2, 4, 6 and 8 weeks of use
  The efficacy variables that will be measured and compared at each time point are:
  Apnea Hypopnea Index (AHI; the number of apneas and hypopneas per hour), mask leak, number of hours of use per night, and user compliance will be measured

OTHER OUTCOMES:
Measure and compare mask performance over a period of 8 weeks | after 2, 4, 6 and 8 weeks of use
  Mask performance will be subjectively assessed by the user over a period of 8 weeks.
  Varibles which will be measured are:
  1. Comfort
  2. Mask seal
  3. Mask stability
  4. The occurence of red marks

CONTACTS AND LOCATIONS:
Locations (1):
- ResMed Ltd, Bella Vista, New South Wales, Australia